CLINICAL TRIAL: NCT00114816
Title: A Randomized Phase III Study Comparing Docetaxel Followed by Cyclophosphamide, Epirubicin and 5-FU to Docetaxel With Capecitabine Followed by Cyclophosphamide, Epirubicin and Capecitabine as Adjuvant Treatment for Early Breast Cancer
Brief Title: Docetaxel Followed by CEF (Cyclophosphamide, Epirubicin and 5-Fluorouracil) Compared to Docetaxel and Capecitabine Followed by CEX (Cyclophosphamide, Epirubicin and Capecitabine) as Adjuvant Treatment for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finnish Breast Cancer Group (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry); AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBCG Protocol No. 01-2003; Roche protocol number MO17728
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; adjuvant; capecitabine; docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel

INTERVENTIONS:
Drug: capecitabine
Drug: docetaxel

SUMMARY:
This study compares two chemotherapy regimens as adjuvant treatment for breast cancer. The study participants are randomly allocated to receive either 3 cycles of docetaxel followed by 3 cycles of CEF (cyclophosphamide, epirubicin and 5-fluorouracil) or to receive 3 cycles of docetaxel plus capecitabine followed by 3 cycles of CEX (cyclophosphamide, epirubicin and capecitabine). The study participants are required to to have a medium to high risk for breast cancer recurrence. The primary aim of the study is to investigate whether addition of capecitabine to a standard taxane/anthracycline regimen will influence recurrence-free survival.

DETAILED DESCRIPTION:
This is an open-label, two-arm, randomized multi-center phase III trial to compare efficacy and safety of a taxane-anthracycline regimen to a taxane-anthracycline-capecitabine regimen as adjuvant treatment of early breast cancer with an intermediate-to-high risk of cancer recurrence.

Patients diagnosed with early breast cancer with an estimated risk of 25% or greater for distant recurrence within 5 years from the diagnosis will be randomly allocated to one of the following 2 arms (1:1):

* Arm A -- 3 cycles of docetaxel 80 mg/m² intravenous (i.v.) (repeated on day [d.] 22); followed by 3 cycles of CEF (cyclophosphamide 600 mg/m2 i.v., epirubicin 75mg/m² i.v., 5-fluorouracil 600 mg/m2 i.v., repeated on d. 22)
* Arm B -- 3 cycles of TX (docetaxel 60 mg/m² i.v., capecitabine twice daily 900 mg/m² given orally on days 1-15 of the cycle; cycle repeated on d. 22); followed by 3 cycles of CEX (cyclophosphamide 600 mg/m2 i.v., epirubicin 75mg/m² i.v, capecitabine twice daily 900 mg/m² on days 1-15 of the cycle; cycle repeated on d. 22)

Locoregional radiotherapy is given according to the institutional practice after completing adjuvant chemotherapy (Tx3/CEFx3 or TXx3/CEXx3).

All patients with ER and/or PgR positive disease will receive adjuvant endocrine therapy. This will consist of 1 mg p.o. anastrozole (ArimidexR) given for 60 months in women who were post-menopausal prior to chemotherapy (no menstrual periods for > 6 months) or of tamoxifen 20 mg p.o. for 60 months in women who were pre-menopausal prior to chemotherapy.

Use of trastuzumab is allowed in HER-2 positive disease.

Patients will be followed up for 5 years post-randomization.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in the study, each patient must fulfill each of the criteria below.

* Have provided written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Be female and 18 years of age or older.
* Have histologically confirmed invasive breast cancer.
* High risk of breast cancer recurrence (> 25% within the first 5 years without adjuvant therapy, > 35% within the first 10 years) with one of the following:

  * Regional node positive disease (pN+; tumor cells or tumor cell clusters < 0.2 mm in diameter are not counted as metastases);
  * Pathological N0 and PgR- and tumor size > 20 mm.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

* > 65 years of age.
* "Special type" histology (mucinous, papillary, medullary, or tubular breast cancer), when pN0.
* ER, PgR and HER-2 status (via in situ hybridization or immunohistochemistry) not determined.
* Presence of distant metastases.
* Previous chemotherapy in the neoadjuvant setting.
* Non-ambulatory or WHO performance status > 1.
* Pregnant or lactating women. Women of childbearing potential (menstruating within 6 months of study entry or with no hysterectomy and age < 55) with either a positive or no pregnancy test at baseline.
* Women of childbearing potential unless using a reliable and appropriate contraceptive method. (Post-menopausal women must have been amenorrheic for at least 6 months to be considered of non-childbearing potential).
* More than 12 weeks between breast surgery and date of randomization.
* Organ allografts with immunosuppressive therapy required.
* Major surgery (except breast surgery) within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* Participation in any investigational drug study within 4 weeks preceding treatment start.
* Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin or carcinoma in situ of the uterine cervix.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 12 months.
* Abnormal laboratory values:

  * Hemoglobin < 10.0 g/dL, neutrophils < 1.5 x 10^9/L, platelet count < 120 x 10^9/L;
  * Serum creatinine > 1.5 x Upper Limit of Normal (ULN);
  * Creatinine clearance (calculated per Cockroft and Gault) < 50 mL/min;
  * Serum bilirubin > ULN;
  * ALAT > 1.5 x ULN;
  * Alkaline phosphatase > 2.5 x ULN.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Lack of physical integrity of the upper gastrointestinal tract or those who have clinically significant malabsorption syndrome.
* Inability to swallow tablets.
* Life expectancy of less than 3 months.
* Unwilling or unable to comply with the protocol for the duration of the study.
* Requirement for concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival

SECONDARY OUTCOMES:
Adverse event rate (CTCAE v. 3.0)
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Heikki T Joensuu, M.D., prof., Principal Investigator — Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland
Locations (1):
- Department of Oncology, Helsinki University Central Hospital, Finland, Helsinki, Finland

REFERENCES:
- [Derived] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola A, Tanner M, Ahlgren J, Auvinen P, Lahdenpera O, Villman K, Nyandoto P, Nilsson G, Poikonen-Saksela P, Kataja V, Bono P, Junnila J, Lindman H. Adjuvant Capecitabine for Early Breast Cancer: 15-Year Overall Survival Results From a Randomized Trial. J Clin Oncol. 2022 Apr 1;40(10):1051-1058. doi: 10.1200/JCO.21.02054. Epub 2022 Jan 12. PMID 35020465
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola-Vuorinen A, Tanner M, Kokko R, Ahlgren J, Auvinen P, Lahdenpera O, Kosonen S, Villman K, Nyandoto P, Nilsson G, Poikonen-Saksela P, Kataja V, Junnila J, Bono P, Lindman H. Adjuvant Capecitabine in Combination With Docetaxel, Epirubicin, and Cyclophosphamide for Early Breast Cancer: The Randomized Clinical FinXX Trial. JAMA Oncol. 2017 Jun 1;3(6):793-800. doi: 10.1001/jamaoncol.2016.6120. PMID 28253390
- [Derived] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola-Vuorinen A, Tanner M, Asola R, Kokko R, Ahlgren J, Auvinen P, Hemminki A, Paija O, Helle L, Nuortio L, Villman K, Nilsson G, Lahtela SL, Lehtio K, Pajunen M, Poikonen P, Nyandoto P, Kataja V, Bono P, Leinonen M, Lindman H; FinXX Study Investigators. Adjuvant capecitabine in combination with docetaxel and cyclophosphamide plus epirubicin for breast cancer: an open-label, randomised controlled trial. Lancet Oncol. 2009 Dec;10(12):1145-51. doi: 10.1016/S1470-2045(09)70307-9. Epub 2009 Nov 10. PMID 19906561